CLINICAL TRIAL: NCT05036096
Title: Cone Beam Breast CT for Breast Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koning Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021SCR
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: Two groups of patients:
  Screening: patients who are scheduled for annual breast cancer screening. Diagnostic: patients who have an abnormality detected by Breast Self Exam, or Clinical Breast Exam (CBE), or have an abnormality detected by an imaging modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CBBCT Imaging Screening Patients (Experimental): Patient undergo bilateral CBBCT imaging (or unilateral CBBCT imaging if the patient had mastectomy) within 4 weeks of screening mammography.
  Interventions: Device: CBBCT Imaging; Device: Digital Mammography
- CBBCT Imaging Diagnostic Patients (Experimental): Patient undergo bilateral CBBCT imaging (or unilateral CBBCT imaging if the patient had mastectomy) within 4 weeks of diagnostic mammography.
  Interventions: Device: CBBCT Imaging; Device: Digital Mammography

INTERVENTIONS:
Device: CBBCT Imaging — Both breasts will be scanned by CBBCT. Only one breast will be scanned if the patient had mastectomy.
Device: Digital Mammography — Both breasts will take digital mammography standard views (CC, MLO) Only one breast will take digital mammography standard views if the patient had mastectomy.

SUMMARY:
Up to one thousand and twenty-eight (1028) patients from screening and diagnostic population will be enrolled and consented to participate in the study to create an enriched data set. These women will be enrolled from annual screening population and diagnostic workup population. The enrolled patient will undergo KBCT scans within 4 weeks of her screening or diagnostic mammography exam and before breast biopsy occurs if biopsy is needed.

DETAILED DESCRIPTION:
Up to one thousand and twenty-eight (1028) patients from screening and diagnostic population will be enrolled and consented to participate in the study to create an enriched data set. These women will be enrolled from annual screening population and diagnostic workup population. The enrolled patient will undergo KBCT scans within 4 weeks of her screening or diagnostic mammography exam and before breast biopsy occurs if biopsy is needed.

Only women will be recruited for this study. Although men can get breast cancer, male breast cancer incidence is low and is not considered to be a great health issue. Thus, this study will exclude males with breast disease.

Women of ages 40 and above will be recruited for participation in the study. There are no enrollment restrictions based on race or ethnic origin. Patients enrolled in the study will have their standard-of-care screening mammography exams performed at the facility. A radiologic technologist, registered in radiography and mammography through the ARRT will perform the Screening Mammography procedure.

For patients enrolled in the study, a bilateral KBCT scan of both breasts (or unilateral scan if the subject has had a mastectomy) will be performed within 4 weeks of the mammography exam.

For all the subjects, the mammograms will be obtained as part of the standard of care and only the 3D KBCT imaging represents additional x-ray exposure.

The KBCT system employs a horizontally oriented gantry beneath a subject support table, which incorporates an x-ray tube at one end and a high-resolution, real-time flat panel detector (FPD) at the opposite end. The system is designed and built-in compliance with the national and international safety standards for medical equipment. A radiologic technologist, registered in radiography and mammography through the ARRT and who is also trained in KBCT acquisition, will position the breast and acquire the images.

For a KBCT scan, the subject lies prone on the support table. The breast of interest is placed through the opening in the table and the breast is positioned in the imaging field. The table sits above a motorized scanning arm carrying an x-ray source and image detector that allows a 360° rotational x-ray sequence in seconds. To acquire the full-volume scan of the breast, the KBCT gantry rotates 360o around the subject's breast, acquiring multiple pulsed projection images. Acquired image data is sent to a computer to perform 3D reconstruction. Specialized 3D visualization software constructs a three-dimensional model of the breast from the images taken during the rotational x-ray sequence. Once the data is reconstructed, it provides 3D isotropic images with the voxel size of ~(0.2mm)3 - ~(0.3mm)3 .The images can be displayed in any plane as well as a 3D rendering.

Our previous studies to-date has illustrated the capacity of the non-contrast KBCT to image the breast without structure overlap and with superior contrast resolution as compared with standard mammography imaging. The study results illustrate that the KBCT system is able to image the entire breast from axillary region to chest wall with clinically acceptable image quality and radiation dose comparable to conventional mammography. Cancers are better visualized as well as defined. In general, it is observed, that cancerous tissues absorb more x-rays than normal tissues, as determined by a higher Hounsfield Unit, but the Hounsfield Unit of some benign lesions can match that of cancer.

The KBCT images will be reviewed by the radiologists who join the study at each site. The radiologist will read the KBCT images and rate each case with "No Recall", "Recall" based on suspicious findings in the images.

ELIGIBILITY:
Inclusion Criteria:

Screening Group:

* Female sex of any ethnicity
* Age 40 years or older
* Scheduled for a routine screening mammography exam within 4 weeks.

Diagnostic Group:

* Female sex of any ethnicity
* Age 30 years or older
* Have an abnormality detected by Breast Self Exam (BSE), or Clinical Breast Exam (CBE), or have an abnormality detected by an imaging modality.
* Will undergo diagnostic mammography, prior to breast biopsy (if needed).

Exclusion Criteria:

* Pregnancy
* Lactation
* Unknown pregnancy status AND

  * has refused pregnancy testing and
  * has refused to sign a pregnancy test waiver
* Women who are unable or unwilling to understand or to provide informed consent
* Women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Women who are unable to tolerate study constraints.
* Women who have received radiation treatments to the thorax or breast area for malignant and nonmalignant conditions, such as (but not limited to):

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkin's disease
* Women who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Women who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to):

  * Tuberculosis
  * Severe scoliosis Additional exclusion criteria due to machine limitations
* Patient's body weight is over the limit of the scanner table (440 lbs. or 200kg)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1024 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiation Dose | 3 months after the CBBCT imaging and Mammography imaging
  The radiation dose of CBBCT imaging and Mammography imaging
Recall Rates | 3 months after CBBCT image review and Mammography image review
  The overall recall rates of CBBCT imaging and Mammography imaging

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Zhang, Ph.D., Study Director — Koning Corporation
Locations (4):
- United States (4):
  - Port Orange Imaging Center, Port Orange, Florida
  - Women's Imaging Specialists, Dacula, Georgia
  - The Howard Center for Women's Health, Tifton, Georgia
  - Knoxville Comprehensive Breast Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No